CLINICAL TRIAL: NCT03923764
Title: Effects of a Diet High in Protein and Energy in Combination With Physical Activity for the Improvement of Coughing Capacity in COPD Patients
Brief Title: High Protein and Energy Diet for Better Coughing in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KOL1
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 1.3 g protein per kg bodyweight per day for 8 weeks
  Interventions: Dietary Supplement: High protein and energy diet
- Kontrol group (Active Comparator): habitual diet
  Interventions: Other: Habitual Diet

INTERVENTIONS:
Dietary Supplement: High protein and energy diet — Intervention group receives nutritional counseling to increase protein and energy in their diet to reach their estimated protein need (1.3 g/kg). Kontrol group continues their usual diet.
  Arms: Intervention group
Other: Habitual Diet — Patients continue their usual diet
  Arms: Kontrol group

SUMMARY:
Chronic Obstructive Lung Disease (COPD) is one of the leading death causes worldwide. COPD is a disease that is characterized by chronic inflammation which leads to irreversible damage of airways and lung tissue. This intervention investigates the effects of a diet high in protein and energy for the improvement of coughing capacity and lung function of COPD patients. The patients will be recruited as part of a lung rehabilitating programme which takes place in Bispebjerg and Hvidovre Hospital. The intervention group receives individual nutritional guidelines whereas the control group continues their usual diet. Blood tests will be performed at baseline and the end of the study. Other anthropometric measures include spirometry for lung function, hand grip strength and fat free mass to assess muscle waisting.

DETAILED DESCRIPTION:
40 patients with COPD randomized to diet with protein 1.3 g/kg/day or habitual intake:

Primary endpoint (before-after): Leicester Cough Questionnaire Secondary endpoints: ADL-score, no. daily cough periods, development in FEV1 and FVC, hand-grib-strenght, use of respiratory medications, smoking, appetite, admissions to hospital, antibiotics and/or steroids, oxygen saturation, FFM (BIA), Coughs tests in spirometer and peak-flow-meter

Study period: 2 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD
* Participating in ongoing lung rehabilitating programme at Hvidovre and Bispebjerg Hospital
* over 18 years

Exclusion Criteria:

* Plasma creatinin over 200 mikrog/l
* dementia
* unable to read or speak danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of coughing capacity of COPD patients | 8 weeks
  Measured by a validated danish version of Leicester Cough Questionnaire (1-7 points)

SECONDARY OUTCOMES:
Weight change | 8 weeks
  kg difference
Oxygen saturation before and after treatment | 8 weeks
  Finger tip measurement - % of normal

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD, MPA, Principal Investigator — Associate Professor
Locations (1):
- Department of Pulmonary Medicine, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No